CLINICAL TRIAL: NCT02397187
Title: The Assessment of the Efficacy of a Structured, Dimension-based, STI (Short Term Intervention) in De-compensated Personality-disorder, Hospitalized, Patients
Brief Title: Efficacy of a Structured, Dimension-based, STI in De-compensated Personality-disorder, Hospitalized, Patients
Acronym: LOOP-PersDis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0003-15-SHA
Record Dates: First submitted 2015-03-05; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Personality Disorders
MeSH Terms: conditions — Personality Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LOOP intervention (Experimental): Patients enrolled in this arm will be treated by the LOOP interventional technique.
  The LOOP conceptualizes the psyche by a three-dimension structure: the space (the potential of experiencing, the "place" where our experiences occur), the content (the experiences themselves; action, thoughts, feelings, experiences and being) and the order (the relationship between the various contents). The LOOP intervene with these three dimensions by a structures scheme, aimed at allowing the patient to quickly reclaim the responsibility on his psyche, stabilize and initiate long-term rehabilitation processes.
  Interventions: Behavioral: LOOP
- TAU (Active Comparator): Patients enrolled in this arm will be TAU, which is based upon short-term supportive PT.
  Interventions: Behavioral: LOOP

INTERVENTIONS:
Behavioral: LOOP — The LOOP conceptualizes the psyche by a three-dimension structure: the space (the potential of experiencing, the "place" where our experiences occur), the content (the experiences themselves; action, thoughts, feelings, experiences and being) and the order (the relationship between the various contents). The LOOP intervene with these three dimensions by a structures scheme, aimed at allowing the patient to quickly reclaim the responsibility on his psyche, stabilize and initiate long-term rehabilitation processes.
  Other Names: ST-CBT / Narrative

SUMMARY:
The assessment of the efficacy of a structured, dimension-based, STI (Short Term Intervention) in de-compensated Personality-disorder, hospitalized, patients

DETAILED DESCRIPTION:
The current study attempts to design a short-term intervention aimed at stabilizing decompensate personality disorder patients in hospitalization. The study is structured as a pilot study, thus will enroll 20 patients only. Patients, upon being hospitalized and after signing the consent to participate in the study, will be randomized to two groups: The first will be treated by the novel, LOOP, concept' the other will be TAU, as routinely done with PersDis patients in the investigators facility. The outcome parameters will be changes in series of questionnaires filled upon being enrolled and at the end of the intervention. Another outcome parameter will be readmission rates in the post-intervention period (3 months).

The LOOP conceptualizes the psyche by a three-dimension structure: the space (the potential of experiencing, the "place" where the investigators experiences occur), the content (the experiences themselves; action, thoughts, feelings, experiences and being) and the order (the relationship between the various contents). The LOOP intervene with these three dimensions by a structures scheme, aimed at allowing the patient to quickly reclaim the responsibility on his psyche, stabilize and initiate long-term rehabilitation processes.

ELIGIBILITY:
Inclusion Criteria:

* Cluster 2 diagnosis
* No suicide attemts 1 month prior to admission
* Regularly treated
* An active support system
* No urgent need for Rx changes

Exclusion Criteria:

* Drug abuse
* An active Axis 1 diagnosis that requires change in Rx
* Unable to read/write fluently

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Questionnaires | up to 28 days
  Questionnaires filled upon being enrolled and at the end of the intervention
Readmission rates | 3 months
  Readmission rates in the post-intervention period (3 months).